CLINICAL TRIAL: NCT04506996
Title: Monday-Focused Tailored Rapid Interactive Mobile Messaging for Weight Management 2
Acronym: M-TRIMM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00007115
Record Dates: First submitted 2020-08-07; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Obesity; Weight Loss; mHealth; Healthy Diet
Keywords: obesity; mHealth; text messages; weight loss intervention; physical activity; diet
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel, superiority randomized controlled trial
Who Masked: Investigator
Masking Description: Participants were randomized after they completed the study's baseline assessment. The randomization sequence was designed to balance treatment groups by gender of the participants. Allocation was concealed from the data collectors, and was determined using a randomization module in REDCap, a survey website. The data collectors were not blinded to the randomization results after the completion of the baseline survey.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - Receiving Text Messages (Experimental): The 16-weeks text-messaging intervention centered around 8 goal topics: eating only when hungry, increasing PA, eating a lower fat diet, eating less sugar and reducing calories from beverages, exercising more, eating a balance diet, portion control, and making healthier food choices in social situations.
  Messaging
  Sun evening: asked to pick 1 of 3 goal topics
  Mon morning: received a goal to focus on for the week
  Mon evening: asked whether plans were made to reach the goal
  Wed morning: received a tip to help reach goal
  Wed evening: reminded that if having cravings, text "tip" to automatically receive a tip
  Fri morning: received end of the week congratulations, encouragement to keep goals in mind over the weekend
  Fri evening: asked for weight, congratulated if lost weight, or encouraged if no weight lost
  Interventions: Behavioral: Monday-Focused Tailored Rapid Interactive Mobile Messaging for Weight Management; Behavioral: Educational Materials
- Control Group - Written Messages (Active Comparator): Participants in the control group, received a printed copy of the same messages that the intervention group received. However, the first eight-weeks' worth of messages and craving tips were given after the baseline assessment, and the rest were given after the first follow-up assessment (~ 8 weeks post randomization).
  The messages for each week were clearly laid out and labeled. Participants were given spaces to record their answers (i.e. to which goal they were selecting for each week). The study staff reviewed the first week's messages together with the study participants to get the participants comfortable with the format that the printed messages were presented in.
  Interventions: Behavioral: Monday-Focused Written Messages for Weight Management; Behavioral: Educational Materials

INTERVENTIONS:
Behavioral: Monday-Focused Tailored Rapid Interactive Mobile Messaging for Weight Management — see arm/group descriptions
  Arms: Intervention Group - Receiving Text Messages
Behavioral: Monday-Focused Written Messages for Weight Management — see arm/group descriptions
  Arms: Control Group - Written Messages
Behavioral: Educational Materials — After the baseline assessment and the 1st follow-up (~8 weeks post randomization), participants received educational materials regarding physical activity and healthier diets. The study staff reviewed these materials with the participants

SUMMARY:
This study, involves the implementation and evaluation of a Monday-focused, individually tailored mobile health application to assist overweight or obese adults who would like to achieve a healthful weight. The goal was to evaluate the application of a Monday-focused delivery system for the M-TRIMM2 intervention on participants who worked or lived in areas in or adjacent to Johns Hopkins East Baltimore medical campus.Targeting mobile messaging occurred at strategic intervals throughout each week, with the intent of prompting participants to renew their health resolutions each Monday combined with lifestyle behavioral education.

DETAILED DESCRIPTION:
The specific aims of this research project are to:

1. Develop a targeted delivery system for mobile health messages which focused on improving physical activity and diet, and setting healthy resolutions each week.
2. Deliver the M-TRIMM intervention, which encourages healthy behavior and the weekly renewal of health resolutions.
3. Evaluate the effectiveness of this intervention on individuals' weight loss, self-efficacy, and motivation to sustain changes in lifestyle behaviors.
4. Assess the benefit of receiving the message content only (in a paper document), versus a scheduled weekly delivery via mobile messaging.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 and <71
* BMI > 25
* having a phone that was capable of receiving text-messages and being willing to receive text-messages

Exclusion Criteria:

* age <18 or ≥ 71
* BMI ≤ 25
* not having a phone that was capable of receiving text-messages or not being willing to receive text-messages

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Percent change in weight from baseline | ~8 weeks, ~16 weeks, and ~42 weeks post-randomization

SECONDARY OUTCOMES:
Body Mass Index (BMI) change from baseline | ~8 weeks, ~16 weeks, and ~42 weeks post-randomization
  BMI = kg/m2

OTHER OUTCOMES:
Change from baseline in self-efficacy to lose weight | ~8 weeks, ~16 weeks, and ~42 weeks post-randomization compared to baseline
  Weight Efficacy Lifestyle Questionnaire (Clark, Abrams,& Niaura, 1991)
Physical activity change from baseline | ~8 weeks, ~16 weeks, and ~42 weeks post-randomization compared to baseline
  International Physical Activity Questionnaire - was used to calculate the total metabolic equivalents (MET)-minutes per week, and MET-minutes per week for four domains of physical activity: (1) PA activity performed at work or during volunteer activities, (2) transportation-related PA (such as walking to do errands), (3) PA performed during housework and caring for family, and (4) recreational, sport, and leisure-time PA.
Change from baseline in fruit and vegetable servings intake from baseline | ~8 weeks, ~16 weeks, and ~42 weeks post-randomization compared to baseline
  National Cancer Institute's (NCI) 19-item All -Day Fruit and Vegetable Screener was used to calculate daily averages of fruit and vegetable serving intake, using NCI's 2001 scoring protocol.
Change from baseline in percent energy from fat intake | ~8 weeks, ~16 weeks, and ~42 weeks post-randomization compared to baseline
  National Cancer Institute's 17-item Percent Energy from Fat Screener - All-Day Quick Food Scan was used and scored according to NCI's 2004 protocol.
Change from baseline in scores of perceived exercise benefits and barriers to engaging in exercise and physical activity | ~8 weeks, ~16 weeks, and ~42 weeks post-randomization compared to baseline
  The 43-item Exercise Benefits and Barriers Scale was used. Separate scores will be calculated for perceived benefits and for perceived barriers. (Sechrist, Walker, & Pender, 1987)
Comparison of satisfaction with the program and suggestions for improvement between intervention and control groups | ~16 weeks, and ~42 weeks post-randomization compared to baseline
  Participants completed a questionnaire that included quantitative and qualitative questions.
  Most of the qualitative questions sought to assess what parts of the program worked well and what could have been done better. For instance, participants were asked for their suggestions about what could be done to improve the M-TRIMM2 program, what messages they liked and did not like, and why they would or would not recommend the program to their friends.
  The quantitative questions covered a variety of topics, including participants engagement with the program (i.e. whether the participants read the messages they received), how useful messages were in helping participants reach the eight study goals (i.e. eating only when hungry, and exercising more), how helpful the goals were helping participants to achieve weight loss, and whether the program helped participants commit to new goals each Monday during the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Cheskin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kharmats AY, Wang C, Fuentes L, Hu L, Kline T, Welding K, Cheskin LJ. Monday-focused tailored rapid interactive mobile messaging for weight management 2 (MTRIMM2): results from a randomized controlled trial. Mhealth. 2022 Jan 20;8:1. doi: 10.21037/mhealth-21-3. eCollection 2022. PMID 35178432